CLINICAL TRIAL: NCT06805201
Title: The Acute Metabolic Impacts of Kaempferia Parviflora Extract in Healthy Men: a Randomized Double Blind Proof of Concept Study
Brief Title: The Effects of Gyngerlean Supplementation on Energy Expenditure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Responsible Party: Principal Investigator, Cassandra Evans, co-investigator, Nova Southeastern University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB 2024-319
Record Dates: First submitted 2025-01-21; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: No Disease or Condition is Being Studied; Metabolism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplement 1 (Experimental): GyngerLean™ 100 mg
  Interventions: Dietary Supplement: Gyngerlean
- Supplement 2 (Experimental): GyngerLean™ 200 mg
  Interventions: Dietary Supplement: Gyngerlean

INTERVENTIONS:
Dietary Supplement: Gyngerlean — Alpinia galangal (Red Ginger), Kaempferia parviflora (Black Ginger), and Zingiber officinale (Yellow Ginger).

SUMMARY:
The goal of this randomized controlled study is to asses the effects of a ginger containing supplement on energy expenditure and substrate utilization in healthy men. The main questions it aims to answer are"

* The effects of Kaempferia parviflora extract on energy expenditure
* The effects of Kaempferia parviflora extract on substrate utilization

ELIGIBILITY:
Inclusion Criteria:

* Active adults. Active is defined as exercising 3 or more times a week for 30 minutes.

Exclusion Criteria:

* Participants must not be diabetics, have Celiac disease, or individuals with pre-existing heart or kidney disease.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-07-23 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2024-08-08 (Actual)

PRIMARY OUTCOMES:
Resting Metabolic rate | 180 minutes
  The amount of energy/calories the body needs to function while at rest.

SECONDARY OUTCOMES:
Respiratory quotient | 180 minutes
  The ratio between carbon dioxide production and oxygen consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Lia Jiannine, Principal Investigator — ljiannine@nova.edu
Locations (1):
- Nova Southeastern University, Davie, Florida, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-28): https://cdn.clinicaltrials.gov/large-docs/01/NCT06805201/Prot_SAP_000.pdf